CLINICAL TRIAL: NCT02007746
Title: Assessment of Liver Fibrosis in Patients With Sickle Cell Disease
Brief Title: Liver Fibrosis in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ofelia Alvarez, Director, Sickle Cell Disease Center, Pediatric Hematology/Oncology, University of Miami
Other Study IDs: 20120222
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; hemochromatosis; liver fibrosis; liver cirrhosis; FibroScan; Ferriscan; liver iron
MeSH Terms: conditions — Anemia, Sickle Cell; Hemochromatosis; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with sickle cell disease and iron overload: Patients will have blood tests done to evaluate liver function and general health, then have FibroScan and Ferriscan. A blinded (no access to laboratory parameters or available data) radiologist will interpret the Ferriscan. Liver biopsy will be also obtained (if not done within the previous year). Otherwise, the results of the recent liver biopsy will be collected.
  Interventions: Other: Liver transient elastography (Fibroscan); Other: Ferriscan; Procedure: Liver biopsy in iron overloaded subjects.
- control patients with sickle cell disease: Patients 10 years and older with sickle cell disease without history of chronic transfusions (less than 4 transfusions in a lifetime) and without obvious liver disease. Will have liver function blood tests and general health check ups. Then will have FibroScan performed. No liver biopsy will be performed in control patients.
  Interventions: Other: Liver transient elastography (Fibroscan)

INTERVENTIONS:
Other: Liver transient elastography (Fibroscan) — Fibroscan will be performed as a measure of liver stiffness. The study will be obtained free of charge in this study.
  Other Names: FibroScan
Other: Ferriscan — Ferriscan will be done to assess the quantity of liver iron in iron overloaded subjects.
  Groups: Subjects with sickle cell disease and iron overload
Procedure: Liver biopsy in iron overloaded subjects. — Liver biopsy will be done and the results will be compared to Fibroscan results.
  Groups: Subjects with sickle cell disease and iron overload

SUMMARY:
Patients with sickle cell disease many have a number of systemic complications, including liver problems. Some of these liver problems lead to liver fibrosis/cirrhosis, secondary to chronic blood transfusions. The purpose of this study is to investigate FibroScan readings in patients with sickle cell disease and iron overload secondary to blood transfusions, and to correlate the FibroScan results with Ferriscan. A comparison with the results of FibroScan to patients with Sickle cell without known liver disease, who have never been on chronic transfusions and with normal liver function profiles will also be made.The primary hypothesis is that the results of FibroScan will correlate with the results of Ferriscan and liver biopsy.

DETAILED DESCRIPTION:
Liver biopsy is the gold standard to examine the liver for iron deposits and histology. However, liver biopsy is invasive and involves a risk of bleeding and pain. Biopsy may also miss significant pathology if the small biopsy specimen is taken from an uninvolved part of the liver. Non-invasive techniques such as MRI are now used to evaluate the liver iron content. MRI can visualize the whole liver and measure liver iron content. MRI, however, will not detect liver scarring.

Liver transient elastography (FibroScan) is a non-invasive ultrasound tool for assessing liver fibrosis or scarring by measuring liver stiffness (LSM). Compared with liver biopsy, FibroScan provides immediate results and is a painless, short (3 mins), simple procedure to perform. In some studies FibroScan reports have correlated well with liver biopsy results of fibrosis and cirrhosis, and with Ferriscan, ferritin and liver function tests.

This purpose of this study is to investigate the role of FibroScan in individuals with sickle cell anemia and iron overload or who have a diagnosis of liver disease, and to compare FibroScan readings with magnetic resonance imaging.

We will also compare the results of the Fibroscan with liver biopsy.

This study will also compare the results of FibroScan to patients with Sickle cell without any known liver disease, who have never been on chronic transfusions (defined as no more than 4 transfusions in lifetime) and who have normal liver function profiles.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients age 10 years and older with sickle cell disease
* meeting other criteria:

  1. history of chronic transfusion and iron overload and/or
  2. known liver disease related to sickle cell or iron overload
* signed consent and assent (as applicable)

Exclusion Criteria:

* children younger than 10 years
* Pregnant females
* Prisoners
* Other causes of liver disease, unrelated to sickle cell or iron overload

Inclusion criteria for controls:

* Patients 10 years and older with sickle cell disease without history of chronic transfusions (less than 4 transfusions in a lifetime)
* and without obvious liver disease.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 30 subjects with sickle cell disease and iron overload. 30 control subjects without history of chronic transfusions (less than 4 transfusions in lifetime) and without evidence of liver pathology.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Liver transient elastography (FibroScan) of liver iron content and stiffness | at imaging visit (3 minutes)
  Liver transient elastography (FibroScan) uses a probe consisting of an ultrasound transducer located at the end of a vibrating piston. The piston produces a vibration of low amplitude and frequency, which generate a shear wave that passes through the skin and liver tissue. The ultrasound then detects the propagation of the shear wave through the liver (at a depth of 25 - 65 mm below the skin surface) by measuring its velocity. The shear wave velocity is directly related to the tissue stiffness, with a higher velocity equating to higher tissue stiffness, corresponding to increasing severity of fibrosis.

SECONDARY OUTCOMES:
magnetic resonance imaging (MRI) measure of liver iron content and stiffness | at imaging visit (about 30-60 minutes)
liver function tests (ALT, AST, serum alkaline phosphate, GGTP, total bilirubin, direct bilirubin), complete blood count, platelets, reticulocyte count, serum ferritin to assess liver function and evaluate overall health | at clinic visit blood draw (about 1 minute)

CONTACTS AND LOCATIONS:
Overall Officials: Ofelia Alvarez, MD, Principal Investigator — University of Miami - Director Sickle Cell Services Pediatric Hematology/Oncology
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Voskaridou E, Plata E, Douskou M, Papadakis M, Delaki EE, Christoulas D, Terpos E. Treatment with deferasirox (Exjade) effectively decreases iron burden in patients with thalassaemia intermedia: results of a pilot study. Br J Haematol. 2010 Jan;148(2):332-4. doi: 10.1111/j.1365-2141.2009.07930.x. Epub 2009 Oct 26. No abstract available. PMID 19863539
- [Result] Fraquelli M, Cassinerio E, Roghi A, Rigamonti C, Casazza G, Colombo M, Massironi S, Conte D, Cappellini MD. Transient elastography in the assessment of liver fibrosis in adult thalassemia patients. Am J Hematol. 2010 Aug;85(8):564-8. doi: 10.1002/ajh.21752. PMID 20658587